CLINICAL TRIAL: NCT01187108
Title: Randomized Controlled Trial of N-acetylcysteine and Acetazolamide in Treatment of Chronic Mountain Sickness
Brief Title: Study of Cobalt's Role in Excessive Erythrocytosis Among High Altitude Dwellers in Cerro de Pasco, Peru
Acronym: CoCMS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other); Jackson, Brian, M.S. (Individual); Thomas H Maren Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-0078
Record Dates: First submitted 2010-08-18; First posted 2010-08-23 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Erythrocytosis; Mountain Sickness
Keywords: Cobalt; Excessive Erythrocytosis; Monge's Disease; Acetazolamide; N-acetylcysteine; Altitude Sickness; Chronic Mountain Sickness
MeSH Terms: conditions — Polycythemia; Altitude Sickness | interventions — Acetylcysteine; Gels; Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo pills (Placebo Comparator)
  Interventions: Drug: Placebo pills
- Acetazolamide alone (Active Comparator)
  Interventions: Drug: Acetazolamide; Drug: Placebo pills
- N-acetylcysteine alone (Active Comparator)
  Interventions: Drug: N-acetylcysteine; Drug: Placebo pills
- Combination of N-acetylcysteine and acetazolamide (Active Comparator)
  Interventions: Drug: N-acetylcysteine; Drug: Acetazolamide

INTERVENTIONS:
Drug: N-acetylcysteine — NAC 600 mg oral once daily
  Other Names: Given in gel capsules
  Arms: Combination of N-acetylcysteine and acetazolamide; N-acetylcysteine alone
Drug: Acetazolamide — Acetazolamide 250 mg oral once daily
  Other Names: Given in gel capsules
  Arms: Acetazolamide alone; Combination of N-acetylcysteine and acetazolamide
Drug: Placebo pills — 1 (or 2 in the placebo group) empty gel capsules
  Arms: Acetazolamide alone; N-acetylcysteine alone; Placebo pills

SUMMARY:
Chronic mountain sickness is characterized by excessive red blood cell production which causes sludging of the vascular system. This high viscosity blood causes heart failure, cognitive dysfunction, and strokes. The investigators hypothesize that cobalt which has been previously been shown to be an environmental pollutant worsens the overproduction of red blood cells. The investigators plan to conduct a 6 week trial in which acetazolamide (already shown to improve chronic mountain sickness) and N-acetylcysteine (a drug that removes cobalt from the blood) are evaluated in their potential to improve chronic mountain sickness.

ELIGIBILITY:
Inclusion Criteria:

* Males over 17 years of age
* Hematocrit > 70%
* Chronic Mountain Sickness score (CMS) > 6
* Able to give informed consent and follow instructions in written Spanish

Exclusion Criteria:

* CMS > 15
* Underlying lung disease, smoking, or oxygen therapy
* Asthma (bronchospasm can be caused by N-acetylcysteine)
* Phlebotomy in last 3 months
* h/o adverse reaction to acetazolamide or N-acetylcysteine

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Hematocrit, or fraction of plasma occupied by cellular elements at week 8 | Baseline and week 8
  Spun hematocrit measured on portable machine

SECONDARY OUTCOMES:
Change from baseline in arterial blood gas values at week 8 | Baseline and week 8
  Analyzed using portable machine. The values analyzed include serum pH, partial pressure of carbon dioxide, partial pressure of oxygen, and serum bicarbonate.
Change from baseline Erythropoietin at week 8 | Baseline and week 8
  Serum hormone that stimulates red blood cell production
Change from baseline in serum and urine Cobalt at day 3 | Baseline and day 3
  Will calculate spot clearance of cobalt
Change in baseline urine protein at 8 weeks | Baseline and week 8
  Ratio of urine total protein to urine creatinine
Change in baseline Chronic mountain sickness score at 8 weeks | Baseline and week 8
  Chronic Mountain Sickness Score Absent Mild Moderate Severe Headache 0 +1 +2 +3 Dizziness 0 +1 +2 +3 Failing Memory 0 +1 +2 +3 Fatigue 0 +1 +2 +3 Breathlessness 0 +1 +2 +3 Sleep disturbances 0 +1 +2 +3 Tinnitus 0 +1 +2 +3 Anorexia 0 +1 +2 +3 Cyanosis of lips, face, or fingers 0 +1 +2 +3 Hyperemia or prominent capillaries conjunctivae or laryngopharynx 0 +1 +2 +3
Changes in baseline Serum electrolytes at day 3, 14 and week 8 | Baseline and Days 3, 14, and week 8
  Electrolytes, specifically monitoring serum potassium to treat serious hypokalemia (serum potassium < 3.0 meQ/L).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Johnson, MD, Principal Investigator — University of Colorado Denver Health Sciences Center; Abdias Hurtado, MD, Principal Investigator — Universidad Peruana Cayetano Heredia; Richard Fuquay, MD, Study Director — University of Colorado Denver Health Sciences Center
Locations (1):
- Chronic mountain sickness clinic, Cerro de Pasco, Departamento de Pasco, Peru

REFERENCES:
- [Background] Jefferson JA, Escudero E, Hurtado ME, Pando J, Tapia R, Swenson ER, Prchal J, Schreiner GF, Schoene RB, Hurtado A, Johnson RJ. Excessive erythrocytosis, chronic mountain sickness, and serum cobalt levels. Lancet. 2002 Feb 2;359(9304):407-8. doi: 10.1016/s0140-6736(02)07594-3. PMID 11844517
- [Background] Jefferson JA, Escudero E, Hurtado ME, Kelly JP, Swenson ER, Wener MH, Burnier M, Maillard M, Schreiner GF, Schoene RB, Hurtado A, Johnson RJ. Hyperuricemia, hypertension, and proteinuria associated with high-altitude polycythemia. Am J Kidney Dis. 2002 Jun;39(6):1135-42. doi: 10.1053/ajkd.2002.33380. PMID 12046023
- [Background] Richalet JP, Rivera-Ch M, Maignan M, Privat C, Pham I, Macarlupu JL, Petitjean O, Leon-Velarde F. Acetazolamide for Monge's disease: efficiency and tolerance of 6-month treatment. Am J Respir Crit Care Med. 2008 Jun 15;177(12):1370-6. doi: 10.1164/rccm.200802-196OC. Epub 2008 Apr 3. PMID 18388356